CLINICAL TRIAL: NCT03817424
Title: A Phase 1 Randomized, Placebo-Controlled, Blinded, Multiple Ascending Dose Study to Evaluate VIB7734 in Systemic Lupus Erythematosus, Cutaneous Lupus Erythematosus, Sjogren's Syndrome, Systemic Sclerosis, Polymyositis, and Dermatomyositis
Brief Title: A Study to Evaluate VIB7734 in Participants With Systemic Lupus Erythematosus (SLE), Cutaneous Lupus Erythematosus (CLE), Sjogren's Syndrome, Systemic Sclerosis, Polymyositis, and Dermatomyositis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: VIB7734.P1b.S1; 2018-003767-60 (EudraCT Number)
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Systemic Lupus Erythematosus; Cutaneous Lupus Erythematosus; Sjogren's Syndrome; Systemic Sclerosis; Polymyositis; Dermatomyositis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Erythematosus, Cutaneous; Sjogren's Syndrome; Scleroderma, Systemic; Polymyositis; Dermatomyositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: VIB7734 Dose 1 (Experimental): Participants will receive VIB7734 Dose 1 via injection q4w for a total of 3 doses on Days 1, 29, and 57.
  Interventions: Drug: VIB7734
- Cohort 2: VIB7734 Dose 2 (Experimental): Participants will receive VIB7734 Dose 2 via injection q4w for a total of 3 doses on Days 1, 29, and 57.
  Interventions: Drug: VIB7734
- Cohort 3: VIB7734 Dose 3 (Experimental): Participants will receive VIB7734 Dose 3 via injection q4w for a total of 3 doses on Days 1, 29, and 57.
  Interventions: Drug: VIB7734
- Placebo (Placebo Comparator): Participants will receive placebo matching to VIB7734 via injection q4w for a total of 3 doses on Days 1, 29, and 57.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIB7734 — Participants will receive VIB7734 via injection.
  Other Names: MEDI7734
  Arms: Cohort 1: VIB7734 Dose 1; Cohort 2: VIB7734 Dose 2; Cohort 3: VIB7734 Dose 3
Drug: Placebo — Participants will receive placebo matching to VIB7734 via injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of escalating, multiple subcutaneous (SC) doses of VIB7734 in participants with Systemic Lupus Erythematosus (SLE), Cutaneous Lupus Erythematosus (CLE), Sjogren's Syndrome, Systemic Sclerosis, Polymyositis, and Dermatomyositis.

DETAILED DESCRIPTION:
This study will have 3 periods: screening, treatment period, and extended follow-up. The screening period is 28 days. A total of 32 participants will be enrolled in 3 cohorts with 8 participants in Cohort 1, and 12 participants each in Cohorts 2 and 3. In Cohort 1, participants will be randomized in a 3:1 ratio to receive VIB7734 or matching placebo by injection every 4 weeks (q4w) for a total of 3 doses on Days 1, 29, and 57. In Cohorts 2 and 3, participants diagnosed with lupus only will be randomized in a 2:1 ratio to receive VIB7734 or matching placebo by injection q4w for 3 doses on Days 1, 29, and 57. Participants will be followed until at least Day 141. After the Day 141 visit, participants will exit the study if participants meets adequate plasmacytoid dendritic cells (pDCs). If an adequate pDC level does not meet at Day 141 visit, the participant will continue the follow-up for pDC repletion until they meet the protocol defined adequate pDC level or Day 337 visit has been reached.

Study acquired from Horizon in 2024. Originally Viela Bio was the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 through 75 years at the time of screening
* Participants with at least one of the following diagnoses:

  1. Systemic Lupus Erythematosus
  2. Cutaneous lupus erythematosus, including acute CLE, subacute CLE, and discoid lupus erythematosus
  3. Sjogren's syndrome (for Cohort 1 only)
  4. Systemic sclerosis (for Cohort 1 only)
  5. Probable or definite polymyositis (for Cohort 1 only)
  6. Probable or definite dermatomyositis (for Cohort 1 only)
* For Cohorts 2 and 3 only: Participants with CLASI activity score greater than or equal to (>=) 8 at both Visits 1 (screening) and 2 (baseline)
* For Cohorts 2 and 3 only: a skin lesion amenable to punch skin biopsy and willingness of the participant to undergo skin biopsy at two time points
* For Cohorts 2 and 3 only: photographs of skin lesions must be submitted for review to confirm the diagnosis of SLE or CLE with active skin lesions confirmation of the diagnosis by the central reviewer must be received prior to randomization
* Females of childbearing potential and nonsterilized males who are ready to use protocol defined contraception methods

Exclusion Criteria:

* Severe manifestations of the diseases under study that could impact the participant safety
* Known history of a primary immunodeficiency or an underlying condition such as known human immunodeficiency virus (HIV) infection, a positive result for HIV infection, splenectomy, or any underlying condition that predisposes the participant to infection
* At screening, have adequate central laboratory test results: aspartate transaminase greater than (>) 2.5 x upper limit of normal (ULN); alanine transaminase >2.5 x ULN; total bilirubin 1.5 x ULN; total immunoglobulin < 500 gram/decilitre; neutrophil count less than (<) 1,000/μL; platelet count < 85,000/μL; haemoglobin < 10 g/dL; glycosylated haemoglobin > 8 percent (%); total lymphocyte count < 300 cells/mm^3; glomerular filtration rate < 50 mL/min/1.73 m^2; plasmacytoid dendritic cells (pDC) level < 0.02% of peripheral blood mononuclear cells (PBMCs)
* Positive test for chronic hepatitis B infection at screening and for hepatitis C virus antibody
* History of or active tuberculosis (TB), or a positive QuantiFERON®-TB Gold test at screening; a primary immunodeficiency or an underlying condition such as known human immunodeficiency virus (HIV) infection, a positive result for HIV infection per central laboratory; cancer; clinically significant cardiac disease
* Herpes zoster infection within 3 months before randomization and/or any severe herpes virus family infection at any time prior to randomization
* Any acute illness or evidence of clinically significant active infection, such as fever >= 38.0 degrees Celsius (>= 100.5 degrees Fahrenheit) at screening (Visit 1) or Day 1 (Visit 2)
* Cohorts 2 and 3 only: use of Group 1 (super-high potency) or Group 2 (high potency) topical corticosteroids
* Receipt of a live-attenuated vaccine within 4 weeks prior to Day 1
* Cohorts 2 and 3 only: have received changing doses of mycophenolate mofetil, methotrexate, leflunomide, azathioprine, or non-steroidal topical immunosuppressants within 28 days before study Day 1 or changing doses of oral or topical corticosteroids within 14 days before study Day 1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs) | Day 1 up to Day 337
Number of Participants With Adverse Events of Special Interest (AESIs) | Day 1 up to Day 337
Number of Participants With Laboratory Abnormalities Reported as TEAEs | Day 1 up to Day 337
Number of Participants With Vital Sign Abnormalities Reported as TEAEs | Day 1 up to Day 337
Number of Participants With 12-Lead Electrocardiogram Abnormalities Reported as TEAEs | Day 1 up to Day 337

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of VIB7734 Maximum Observed Serum Concentration (Cmax) of VIB7734 | Days 1 (pre-dose), 8, 15, 29 (pre-dose), 36, 43, 57 (pre-dose), 64, 71, 85, 113, 141, 169, 197, 225, and 253
Area Under the Concentration-time Curve (AUC) of VIB7734 | Days 1 (pre-dose), 8, 15, 29 (pre-dose), 36, 43, 57 (pre-dose), 64, 71, 85, 113, 141, 169, 197, 225, and 253
Systemic Clearance (CL) of VIB7734 | Days 1 (pre-dose), 8, 15, 29 (pre-dose), 36, 43, 57 (pre-dose), 64, 71, 85, 113, 141, 169, 197, 225, and 253
Terminal Half-life (t1/2) of VIB7734 | Days 1 (pre-dose), 8, 15, 29 (pre-dose), 36, 43, 57 (pre-dose), 64, 71, 85, 113, 141, 169, 197, 225, and 253
Number of Participants With Positive Anti-Drug Antibodies of VIB7734 | Day 1 up to Day 309
Change from Baseline in Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Activity Score (Cohorts 2 and 3) | Day 1 up to Day 253
Blood Levels of pDCs | Day 1 up to Day 337

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (30):
- United States (19):
  - Viela Bio Investigative Site, Anniston, Alabama
  - Viela Bio Investigative Site, Birmingham, Alabama
  - Viela Bio Investigative Site, Los Angeles, California
  - Viela Bio Investigative Site, Upland, California
  - Viela Bio Investigative Site, Danbury, Connecticut
  - Viela Bio Investigative Site, Fort Lauderdale, Florida
  - Viela Bio Investigative Site, Hialeah, Florida
  - Viela Bio Investigative Site, Jacksonville, Florida
  - Viela Bio Investigative Site, Miami Lakes, Florida
  - Viela Bio Investigative Site, St. Petersburg, Florida
  - Viela Bio Investigative Site, Lawrenceville, Georgia
  - Viela Bio Investigative Site, Great Neck, New York
  - Viela Bio Investigative Site, Charlotte, North Carolina
  - Viela Bio Investigative Site, Durham, North Carolina
  - Viela Bio Investigative Site, Duncansville, Pennsylvania
  - Viela Bio Investigative Site, Philadelphia, Pennsylvania
  - Viela Bio Investigative Site, Memphis, Tennessee
  - Viela Bio Investigative Site, Allen, Texas
  - Viela Bio Investigative Site, Mesquite, Texas
- Poland (7):
  - Viela Bio Investigative Site, Bialystok
  - Viela Bio Investigative Site, Bydgoszcz
  - Viela Bio Investigative Site, Krakow
  - Viela Bio Investigative Site, Poznan
  - Viela Bio Investigative Site, Rzeszów
  - Viela Bio Investigative Site, Warsaw
  - Viela Bio Investigative Site, Wroclaw
- Spain (4):
  - Viela Bio Investigative Site, Barcelona
  - Viela Bio Investigative Site, Bilbao
  - Viela Bio Investigative Site, Madrid
  - Viela Bio Investigative Site, Seville

IPD SHARING:
Plan to Share IPD: No